CLINICAL TRIAL: NCT06431620
Title: Safety and Efficacy of Recombinant Human Thyroid Stimulating Hormone for Adjuvant Diagnosis in Patients With Locally Advanced/Metastatic Differentiated Thyroid Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Feng Wang, Director of nuclear medicine department, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20240514-03
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Recombinant Human Thyroid Stimulating Hormone
MeSH Terms: interventions — Thyrotropin Alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rhTSH group (Experimental): rhTSH is used to raise blood TSH levels to meet the requirements of diagnostic 131I SPECT/CT whole-body scans before and after TKI medication.
  Interventions: Drug: Recombinant Human Thyroid Stimulating Hormone

INTERVENTIONS:
Drug: Recombinant Human Thyroid Stimulating Hormone — recombinant human thyrotropin (rhTSH) injection: 0.9mg/1.0mL/piece; intramuscular injection; once a day for two consecutive days.

SUMMARY:
Exogenous injection of recombinant human thyroid stimulating hormone (rhTSH) can elevate TSH in the short term (2 days) to meet the requirements of diagnostic 131I SPECT/CT whole-body scans. Antiangiogenic tyrosine kinase inhibitors (TKI) couuld alter the uptake of radioactive 131I in locally advanced or metastatic differentiated thyroid cancer. rhTSH can help to perform the diagnostic 131I SPECT/CT whole-body scans before and after the TKI usage. rhTSH can reduce the risk of tumor progression caused by thyroid hormone withdrawal period and the side effects of hypothyroidism also caused by thyroid hormone withdrawal, and clarify the 131I uptake change after TKI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18~75 years old (including 18 and 75 years old);
* ECOG: 0-2 points;
* Expected survival of more than 3 months; Differentiated thyroid carcinoma undergoing total thyroidectomy or subtotal thyroidectomy and confirmed as locally recurrent or metastatic disease by imaging, serum tumor marker (tg), biopsy pathology; at least one measurable lesion (diameter of the tumor ≥10 mm), and meets the requirements of RECIST 1.1.
* Hemoglobin ≥80g/L, neutrophil ≥1.5×109/L, platelet count ≥80×109/L, serum creatinine ≤1.5× upper limit of normal or creatinine clearance ≥60ml/min, Blood urea nitrogen ≤2.5× upper limit of normal (ULN); Total bilirubin ≤1.5×ULN; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN; If accompanied by liver metastasis, ALT and AST≤5×ULN albumin ≥25 g/L;
* Women of childbearing potential must have taken reliable contraceptive measures or undergone a pregnancy test (serum or urine) within 7 days prior to enrollment, with a negative result, and be willing to use appropriate contraceptive methods during the trial and for 1 year after the last dose of 131I (for women), or for 6 months after the last dose of 131I (for men);
* Participants voluntarily joined the study and signed informed consent, with good compliance and follow-up;
* Patients diagnosed with iodine-refractory/potentially iodine-refractory DTC after multidisciplinary team discussion.

Exclusion Criteria:

* Accompanied by pleural effusion or ascites, causing respiratory distress;
* Symptoms of brain metastasis cannot be controlled and treated in less than 2 months; there is a risk of suffocation due to excessively large neck metastatic masses; patients with spinal bone metastases have a risk of spinal cord compression paralysis; cardiac metastasis, heart failure, and patients at risk of acute cardiovascular events;
* Patients with severe and uncontrolled diseases, including: 1) Uncontrolled hypertension (despite optimal drug therapy, systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg); 2) Poorly controlled arrhythmias of ischemic heart disease or myocardial infarction of grade II or above (including corrected QT interval (QTc) male ≥450 ms, female ≥470 ms) and ≥2 congestive heart failures (New York Heart Association (NYHA) classification); 3) Poorly controlled diabetes (fasting blood sugar >10mmol/L); 4) Active or poorly controlled severe infections (according to Common Terminology Criteria for Adverse Events ≥ grade 2); 5) Patients with active hepatitis B or hepatitis C (hepatitis B: positive HBsAg and hepatitis B virus (HBV) DNA ≥500 IU/mL; hepatitis C: positive hepatitis C virus (HCV) RNA and abnormal liver function), or active infections requiring antimicrobial therapy (e.g., with antibiotics, antiviral drugs, antifungal drugs); 6) Renal insufficiency: urine routine shows urine protein ≥++ or confirmed 24-hour urine protein ≥1.0 g; 7) Patients with seizures requiring treatment.
* Received surgical treatment, incisional biopsy, or major trauma within 28 days prior to randomization;
* Unable to quit or with a history of psychiatric medication abuse;
* Allergic to the investigational drug (rhTSH or 131I) or its excipients;
* Had an infection within 4 weeks prior to screening, including bacterial, viral, or fungal infections, with ongoing symptoms at the time of screening;
* Received lipophilic iodine contrast agents (such as iodized oil, iodized benzene, etc.) within the past 3 months or received water-soluble iodine contrast agents (such as iohexol, iodinated glycerol, etc.) within the past 1 month prior to screening;
* Pregnant or lactating women, or women who engaged in unprotected sexual intercourse within the two weeks prior to screening, or women with a positive blood pregnancy test at screening;
* Male subjects (or their partners) or female subjects who have plans for fertility or donation of sperm or ova during the entire study period and within 6 months after the end of the study, and who are unwilling to adopt contraceptive measures during the study period and within 6 months after the end of the study;
* Researchers believe that the presence of any condition may harm the subjects or prevent them from meeting or fulfilling the study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
TSH | 24 hours after the second TSH injection
  The proportion of patients with thyroid stimulating hormone>30 mIU/L

SECONDARY OUTCOMES:
Positive diagnosis rate of lesions | 72 hours after 131I treatment until progression or death, whichever came first
  Positive diagnosis rate of lesions in diagnostic 131I SPECT/CT whole-body scans

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical Univerity, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No